CLINICAL TRIAL: NCT03500055
Title: Does Implementation of an Abdominal Closure Bundle in Patients Undergoing Scheduled Cesarean Section Lead to Reduction in Surgical Site Infection? - A Randomized Controlled Trial
Brief Title: Abdominal Closure Bundle to Reduce Surgical Site Infection in Patients Undergoing C-sections. Cesarean Section Lead to Reduction in Surgical Site Infection? - A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abington Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shaina Bruce, Resident physician, Abington Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-016
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Surgical Site Infection; Cesarean Section; Infection
MeSH Terms: conditions — Surgical Wound Infection; Infections

STUDY DESIGN:
Intervention Model Description: Single center, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Only the primary investigators will be able to be blinded for this study. The surgeon is unable to be blinded and since the patient is awake during c-sections, blinding will be impossible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Closure Bundle (Experimental): Surgeons will re-scrub, change gown and gloves prior to closure of fascia. Will also use new instruments, bovie tip, suction tip, and light handles, for closure of fascia, subcutaneous tissue, and skin.
  Interventions: Procedure: Abdominal Closure Bundle
- Control (No Intervention): Normal operative procedure. The abdominal closure bundle will not be used.

INTERVENTIONS:
Procedure: Abdominal Closure Bundle — Surgeons will re-scrub, change gown and gloves prior to closure of fascia. Will also use new instruments, bovie tip, suction tip, and light handles, for closure of fascia, subcutaneous tissue, and skin
  Arms: Abdominal Closure Bundle

SUMMARY:
This study is a single center, randomized controlled trial investigating the use of an abdominal closure bundle to reduce surgical site infection in patients undergoing cesarean section. The abdominal closure bundle consists of surgeon repeat scrub, changing gown and gloves, as well as usage of new instruments for closure of fascia, subcutaneous tissue, and skin. Patients will be randomized to either abdominal closure bundle or normal operative procedure. Primary outcome is surgical site infection within 30 days of procedure.

DETAILED DESCRIPTION:
All patients, aged 18 years or older, greater than 34 weeks of gestation who will be undergoing a scheduled cesarean section to be performed by Abington Primary Women's Health Care Group, Abington Ob/Gyn Associates, Womencare, Women's Health Care Group, Dr. Ron Hoffman, or the Ob/Gyn Chief Service will be considered for participation in this study. Scheduled cesarean sections include all routine cesarean sections- whether receiving spinal or general anesthesia, as well as patients who present to obstetrical triage in labor or with ruptured membranes who are for cesarean section.

The following patients will be excluded from our study:

* Unscheduled, STAT or urgent cesarean sections from the labor floor (failure to descend, failure to progress, non-reassuring fetal heart tracing, chorioamnionitis, placental abruption, prolapsed cord, etc.)
* SOAT (Surgical Operative Assist Team) cesarean sections
* Gestational age < 34 weeks for any reason
* Preterm premature rupture of membranes from antepartum unit

As there are no published prospective trials abdominal closure bundles in cesarean sections, sample size calculations were completed using a recently published meta-analysis of multiple retrospective studies.4 These studies investigated various surgical site reduction techniques as applied to cesarean sections. Using this data, which shows an average pre-intervention SSI rate of 6% and post-reduction SSI rate of 2%, to detect a statistically significant reduction, we will need to enroll approximately 850 patients.

Patients will be randomly assigned to receive either normal operative procedure or the closing bundle through a randomized process. Simple randomization in a 1:1 ratio will be completed via Microsoft Excel. Group assignments will be placed in sealed opaque envelopes which will be located on the labor and delivery unit. The envelope will be opened by the resident physician or advanced practice professional who will be assisting with the cesarean section on arrival to the operating room. This will allow the scrub tech to prepare the closing tray prior to the start of the procedure if indicated.

All patients will receive pre-operative antibiotics, chlorhexidine abdominal preparation, thirty second betadine vaginal preparation, hair removal by clippers at the operative site, lower extremity forced air warmer, subcutaneous tissue closure >2cm, subcuticular skin closure, and removal of surgical bandage on post-operative day 2. The abdominal closure bundle includes changing of the surgical gown and gloves, repeat surgical scrub, and usage of new surgical instruments, light handles, suction, and bovie tip for closure of fascia, subcutaneous tissue, and skin. Given the nature of the intervention, the surgeon and patient will not be blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Greater than 34 weeks of gestation who will be undergoing a scheduled cesarean section to be performed by Abington Primary Women's Health Care Group, Abington Ob/Gyn Associates, Womencare, Women's Health Care Group, Dr. Ron Hoffman, or the Ob/Gyn Chief Service will be considered for participation in this study.
* Patients who present to obstetrical triage in labor or with ruptured membranes who are for cesarean section are also included in the study.

Exclusion Criteria:

* Unscheduled, STAT or urgent cesarean sections from the labor floor (failure to descend, failure to progress, non-reassuring fetal heart tracing, chorioamnionitis, placental abruption, prolapsed cord, etc.)
* SOAT (Surgical Operative Assist Team) cesarean sections
* Gestational age < 34 weeks for any reason
* Preterm premature rupture of membranes from antepartum unit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | Within 30 days of procedure.
  Definitions per 2017 CDC definitions

SECONDARY OUTCOMES:
Risk factors for surgical site infection | Within 30 days of procedure.
  Will collect demographic, obstetrical, and surgical characteristics and determine specific risk factors for surgical site infection in these patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Abington Hospital-Jefferson Health, Abington, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pellegrini JE, Toledo P, Soper DE, Bradford WC, Cruz DA, Levy BS, Lemieux LA. Consensus Bundle on Prevention of Surgical Site Infections After Major Gynecologic Surgery. J Obstet Gynecol Neonatal Nurs. 2017 Jan-Feb;46(1):100-113. doi: 10.1016/j.jogn.2016.10.003. Epub 2016 Dec 8. PMID 27955845
- [Background] Schiavone MB, Moukarzel L, Leong K, Zhou QC, Afonso AM, Iasonos A, Roche KL, Leitao MM Jr, Chi DS, Abu-Rustum NR, Zivanovic O. Surgical site infection reduction bundle in patients with gynecologic cancer undergoing colon surgery. Gynecol Oncol. 2017 Oct;147(1):115-119. doi: 10.1016/j.ygyno.2017.07.010. Epub 2017 Jul 19. PMID 28734498
- [Background] Lachiewicz MP, Moulton LJ, Jaiyeoba O. Pelvic surgical site infections in gynecologic surgery. Infect Dis Obstet Gynecol. 2015;2015:614950. doi: 10.1155/2015/614950. Epub 2015 Feb 18. PMID 25788822
- [Background] Carter EB, Temming LA, Fowler S, Eppes C, Gross G, Srinivas SK, Macones GA, Colditz GA, Tuuli MG. Evidence-Based Bundles and Cesarean Delivery Surgical Site Infections: A Systematic Review and Meta-analysis. Obstet Gynecol. 2017 Oct;130(4):735-746. doi: 10.1097/AOG.0000000000002249. PMID 28885421
- [Background] Bruce SF, Carr DN, Burton ER, Sorosky JI, Shahin MS, Naglak MC, Edelson MI. Implementation of an abdominal closure bundle to reduce surgical site infection in patients on a gynecologic oncology service undergoing exploratory laparotomy. Gynecol Oncol. 2018 Jun;149(3):560-564. doi: 10.1016/j.ygyno.2018.03.045. Epub 2018 Mar 14. PMID 29548786
- See also: 2017 CDC Surgical Site Infection Guidelines — http://www.cdc.gov/nhsn/PDFs/pscManual/9pscSSIcurrent.pdf